CLINICAL TRIAL: NCT04909645
Title: A Comparison of Invasive and Non-invasive Measurement of Cardiac Index and Systemic Vascular Resistance in Living Donor Liver Transplantation
Brief Title: A Comparison of Invasive and Non-invasive Measurement of CI and SVR in Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seong Mi Yang, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2104-037-1209
Record Dates: First submitted 2021-05-10; First posted 2021-06-02 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Living Donor Liver Transplantation
Keywords: finger cuff; systemic vascular resistance; cardiac index; noninvasive monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clearsight (finger cuff) (Experimental)
  Interventions: Diagnostic Test: Clearsight (finger cuff)

INTERVENTIONS:
Diagnostic Test: Clearsight (finger cuff) — Clearsight (Edwards Lifesciences, Irvine, CA), a noninvasive technique, uses a finger cuff to measure blood pressure, cardiac output (CO) and cardiac index. Systemic vascular resistance (SVR) is calculated by the following equation: SVR=(Mean arterial pressure-Central venous pressure)*80/CO.

SUMMARY:
Patients who are scheduled to receive living donor liver transplantation will be monitored with a radial and femoral arterial line. A pulmonary artery catheter will also be placed and central venous pressure, cardiac index, and cardiac output will also be monitored. Simultaneously, on the middle finger of the hand where the radial artery is monitored, Clearsight (Edwards Lifesciences, Irvine, CA), a finger cuff, is placed and noninvasive blood pressure, cardiac output, cardiac index are measured. Using the VitalDB program, the parameters measured with the invasive methods and the parameters obtained by the noninvasive method are compared.

DETAILED DESCRIPTION:
In many end stage liver disease patients, cardiac output (CO) is increased and systemic vascular resistance (SVR) is decreased. During liver transplantation it is common to see hemodynamic instability due to massive blood loss and clamping of the major vessels. As a result invasive monitoring via a pulmonary catheter is usually done to continuously monitor the CO and SVR. However, because of its invasiveness, complications such as pulmonary artery rupture and ventricular arrhythmia can occur.

Clearsight (Edwards Lifesciences, Irvine, CA) is a noninvasive technique using a finger cuff to measure not only blood pressure but also CO and cardiac index (CI).

There have been previous reports on the correlation of this noninvasive method in other patient populations but no studies have been done in liver recipients. Also no studies have been done comparing SVR.

Patients presenting for living donor liver transplantation are anesthetized according to the SNUH protocol. Right radial and femoral arterial lines are placed. A central catheter is placed in the right jugular vein and a pulmonary artery catheter (Swan-Ganz CCOmbo CCO/SvO2™; Edward Lifesciences LLC, Irvine, CA, USA) is placed. This is connected to the Vigilance™ hemodynamic monitor (Edwards Lifesciences) and central venous pressure (CVP), CO, CI are monitored and SVR is calculated by the following equation: SVR=(Mean arterial pressure-CVP)*80/CO. The Clearsight system is connected after the finger cuff is placed on the middle finger of the right hand. Blood pressure, CO, CI are measured and SVR is calculated.

The variables are compared in the following phases:

Phase 1 (preanhepatic1): induction complete (baseline) Phase 2 (preanhepatic2): induction - recipient hepatectomy Phase 3 (anhepatic1): recipient hepatectomy - Inferior Vena Cava (IVC) clamping Phase 4 (anhepatic2): IVC clamping - reperfusion Phase 5 (neohepatic1 [reperfusion]) Reperfusion - 5 minutes postreperfusion Phase 6 (neohepatic2): 20 minutes after reperfusion Phase 7 (neohepatic3): 1 hour after reperfusion

The investigators hypothesize that the noninvasive hemodynamic monitoring method by the Clearsight will be able to replace the invasive monitoring by the pulmonary artery catheter.

ELIGIBILITY:
Inclusion Criteria:

* routine living donor liver transplantation recipients needing pulmonary artery catheterization who have been informed and given consent

Exclusion Criteria:

* Patients with atrial fibrillation
* Contraindications to pulmonary artery catheterization or needing attention to insertion of pulmonary artery catheter: right-sided endocarditis, tumors, right sided valvular disease, left bundle branch block
* Patients with obstructive vascular disease in the upper extremities, anatomical deformities in the upper extremities, Raynaud syndrome, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-05-28 (Estimated); Study Completion 2022-05-28 (Estimated)

PRIMARY OUTCOMES:
comparison of invasive and non-invasive measurement for cardiac index | Phase 1 (preanhepatic1): completion of the anesthetic induction (baseline)
  cardiac index
comparison of invasive and non-invasive measurement for systemic vascular resistance | Phase 1 (preanhepatic1): completion of the anesthetic induction (baseline)
  systemic vascular resistance measured by the following equation: SVR=(Mean arterial pressure-central venous pressure)*80/cardiac output.
  Femoral MAP is used for the invasive measurement
comparison of invasive and non-invasive measurement for cardiac index | Phase 2 (preanhepatic2): 60 minutes after the anesthetic induction
  cardiac index
comparison of invasive and non-invasive measurement for systemic vascular resistance | Phase 2 (preanhepatic2): 60 minutes after the anesthetic induction
  systemic vascular resistance measured by the following equation: SVR=(Mean arterial pressure-central venous pressure)*80/cardiac output.
  Femoral MAP is used for the invasive measurement
comparison of invasive and non-invasive measurement for cardiac index | Phase 3 (anhepatic 1): 10 minutes after recipient hepatectomy is complete
  cardiac index
comparison of invasive and non-invasive measurement for systemic vascular resistance | Phase 3 (anhepatic 1): 10 minutes after recipient hepatectomy is complete
  systemic vascular resistance measured by the following equation: SVR=(Mean arterial pressure-central venous pressure)*80/cardiac output.
  Femoral MAP is used for the invasive measurement
comparison of invasive and non-invasive measurement for cardiac index | Phase 4 (anhepatic 2): 10 minutes after IVC clamping
  cardiac index
comparison of invasive and non-invasive measurement for systemic vascular resistance | Phase 4 (anhepatic 2): 10 minutes after IVC clamping
  systemic vascular resistance measured by the following equation: SVR=(Mean arterial pressure-central venous pressure)*80/cardiac output.
  Femoral MAP is used for the invasive measurement
comparison of invasive and non-invasive measurement for cardiac index | Phase 5 (neohepatic1 [reperfusion]): 5 minutes after reperfusion
  cardiac index
comparison of invasive and non-invasive measurement for systemic vascular resistance | Phase 5 (neohepatic1 [reperfusion]): 5 minutes after reperfusion
  systemic vascular resistance measured by the following equation: SVR=(Mean arterial pressure-central venous pressure)*80/cardiac output.
  Femoral MAP is used for the invasive measurement
comparison of invasive and non-invasive measurement for cardiac index | Phase 6(neohepatic2): 20 minutes after reperfusion
  cardiac index
comparison of invasive and non-invasive measurement for systemic vascular resistance | Phase 6(neohepatic2): 20 minutes after reperfusion
  systemic vascular resistance measured by the following equation: SVR=(Mean arterial pressure-central venous pressure)*80/cardiac output.
  Femoral MAP is used for the invasive measurement
comparison of invasive and non-invasive measurement for cardiac index | Phase 7(neohepatic3): 1 hour after reperfusion
  cardiac index
comparison of invasive and non-invasive measurement for systemic vascular resistance | Phase 7(neohepatic3): 1 hour after reperfusion
  systemic vascular resistance measured by the following equation: SVR=(Mean arterial pressure-central venous pressure)*80/cardiac output.
  Femoral MAP is used for the invasive measurement

SECONDARY OUTCOMES:
comparison of invasive and non-invasive measurement for systolic and diastolic blood pressure | Phase 1 (preanhepatic1): completion of the anesthetic induction (baseline)
  systolic and diastolic blood pressure
comparison of invasive and non-invasive measurement for systolic and diastolic blood pressure | Phase 2 (preanhepatic2): 60 minutes after the anesthetic induction
  systolic and diastolic blood pressure
comparison of invasive and non-invasive measurement for systolic and diastolic blood pressure | Phase 3 (anhepatic 1): 10 minutes after recipient hepatectomy is complete
  systolic and diastolic blood pressure
comparison of invasive and non-invasive measurement for systolic and diastolic blood pressure | Phase 4 (anhepatic 2): 10 minutes after IVC clamping
  systolic and diastolic blood pressure
comparison of invasive and non-invasive measurement for systolic and diastolic blood pressure | Phase 5 (neohepatic1 [reperfusion]): 5 minutes after reperfusion
  systolic and diastolic blood pressure
comparison of invasive and non-invasive measurement for systolic and diastolic blood pressure | Phase 6(neohepatic2): 20 minutes after reperfusion
  systolic and diastolic blood pressure
comparison of invasive and non-invasive measurement for systolic and diastolic blood pressure | Phase 7(neohepatic3): 1 hour after reperfusion
  systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Seong Mi Yang, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Wolf AM. 6/2/06 Perioperative assessment of the cardiovascular system in ESLD and transplantation. Int Anesthesiol Clin. 2006 Fall;44(4):59-78. doi: 10.1097/01.aia.0000210818.85287.de. No abstract available. PMID 17033479
- [Background] Rudnick MR, Marchi LD, Plotkin JS. Hemodynamic monitoring during liver transplantation: A state of the art review. World J Hepatol. 2015 Jun 8;7(10):1302-11. doi: 10.4254/wjh.v7.i10.1302. PMID 26052376
- [Background] Evans DC, Doraiswamy VA, Prosciak MP, Silviera M, Seamon MJ, Rodriguez Funes V, Cipolla J, Wang CF, Kavuturu S, Torigian DA, Cook CH, Lindsey DE, Steinberg SM, Stawicki SP. Complications associated with pulmonary artery catheters: a comprehensive clinical review. Scand J Surg. 2009;98(4):199-208. doi: 10.1177/145749690909800402. PMID 20218415
- [Background] Saugel B, Hoppe P, Nicklas JY, Kouz K, Korner A, Hempel JC, Vos JJ, Schon G, Scheeren TWL. Continuous noninvasive pulse wave analysis using finger cuff technologies for arterial blood pressure and cardiac output monitoring in perioperative and intensive care medicine: a systematic review and meta-analysis. Br J Anaesth. 2020 Jul;125(1):25-37. doi: 10.1016/j.bja.2020.03.013. Epub 2020 May 29. PMID 32475686
- [Background] Saugel B, Cecconi M, Wagner JY, Reuter DA. Noninvasive continuous cardiac output monitoring in perioperative and intensive care medicine. Br J Anaesth. 2015 Apr;114(4):562-75. doi: 10.1093/bja/aeu447. Epub 2015 Jan 16. PMID 25596280
- [Background] Kim SH, Lilot M, Sidhu KS, Rinehart J, Yu Z, Canales C, Cannesson M. Accuracy and precision of continuous noninvasive arterial pressure monitoring compared with invasive arterial pressure: a systematic review and meta-analysis. Anesthesiology. 2014 May;120(5):1080-97. doi: 10.1097/ALN.0000000000000226. PMID 24637618
- [Background] Al-Hamoudi WK. Cardiovascular changes in cirrhosis: pathogenesis and clinical implications. Saudi J Gastroenterol. 2010 Jul-Sep;16(3):145-53. doi: 10.4103/1319-3767.65181. PMID 20616408
- [Background] Kanazawa H, Maeda T, Miyazaki E, Hotta N, Ito S, Ohnishi Y. Accuracy and Trending Ability of Blood Pressure and Cardiac Index Measured by ClearSight System in Patients With Reduced Ejection Fraction. J Cardiothorac Vasc Anesth. 2020 Dec;34(12):3293-3299. doi: 10.1053/j.jvca.2020.03.045. Epub 2020 Apr 20. PMID 32404245
- [Background] Sumiyoshi M, Maeda T, Miyazaki E, Hotta N, Sato H, Hamaguchi E, Kanazawa H, Ohnishi Y, Kamei M. Accuracy of the ClearSight system in patients undergoing abdominal aortic aneurysm surgery. J Anesth. 2019 Jun;33(3):364-371. doi: 10.1007/s00540-019-02632-6. Epub 2019 Mar 23. PMID 30904953
- [Background] Lee HC, Jung CW. Vital Recorder-a free research tool for automatic recording of high-resolution time-synchronised physiological data from multiple anaesthesia devices. Sci Rep. 2018 Jan 24;8(1):1527. doi: 10.1038/s41598-018-20062-4. PMID 29367620
- [Background] Critchley LA, Critchley JA. A meta-analysis of studies using bias and precision statistics to compare cardiac output measurement techniques. J Clin Monit Comput. 1999 Feb;15(2):85-91. doi: 10.1023/a:1009982611386. PMID 12578081
- [Background] Suehiro K, Tanaka K, Funao T, Matsuura T, Mori T, Nishikawa K. Systemic vascular resistance has an impact on the reliability of the Vigileo-FloTrac system in measuring cardiac output and tracking cardiac output changes. Br J Anaesth. 2013 Aug;111(2):170-7. doi: 10.1093/bja/aet022. Epub 2013 Mar 10. PMID 23479677